CLINICAL TRIAL: NCT04346147
Title: Prospective, Phase II, Randomized, Open-label, Parallel Group Study to Evaluate the Efficacy of Baricitinib, Imatinib or Supportive Treatment in Patients With SARS Cov2 Pneumonia
Brief Title: Clinical Trial to Evaluate Efficacy of 3 Types of Treatment in Patients With Pneumonia by COVID-19
Acronym: Covid19COVINIB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario de Fuenlabrada (Other)
Collaborators: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24032020
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Imatinib Mesylate; baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Imatinib 400 mg (Experimental): Imatinib 400 mg 1 tablet 24 hours
  Interventions: Drug: Imatinib tablets
- Baricitinib 4 mg (Experimental): Baricitinib 4 mg 1 tablet 24 hours
  Interventions: Drug: Baricitinib Oral Tablet
- Supportive treatment (Experimental): Any therapeutic intervention aimed at the control of clinical deterioration is contemplated without initiating or having previously initiated any drug with potential beneficial effect previously described in vitro or in pre-clinical / clinical models against SARS-CoV-2 prior to patient recruitment.
  Interventions: Other: Supportive tratment

INTERVENTIONS:
Drug: Imatinib tablets — Imatinib 400 mg QD oral
  Other Names: Arm A
  Arms: Imatinib 400 mg
Drug: Baricitinib Oral Tablet — Baricitinib 4 mg QD oral
  Other Names: Arm B
  Arms: Baricitinib 4 mg
Other: Supportive tratment — Any therapeutic intervention aimed at the control of clinical deterioration is contemplated without initiating or having previously initiated any drug with potential beneficial effect previously described in vitro or in pre-clinical / clinical models against SARS-CoV-2 prior to patient recruitment.
  Other Names: Best care
  Arms: Supportive treatment

SUMMARY:
In absence of vaccine and medications specifically designed to treat SARS-CoV-2 disease, identifying treatment options is critical at this time to control the disease outbreak.

For this, we have designed a phase II trial of efficacy and safety with 3 branches of different combinations of treatment to identify which is the best early treatment option for patients with pneumonia due to SARS-CoV-2 (Covid-19) Identifying treatment options as early as possible is critical to the SARS-CoV-2 outbreak response. Currently, there is no approved vaccine for the disease and the treatments being used are not specifically designed for the SARS-CoV-2 virus, but are different groups of drugs used for other pathologies with mechanisms of action that justify their use because they inhibit entry of the virus into virus cells or proteases.

The study aims to compare Imatinib 400mg, Baricitinib 4mg or supportive treatment, administered for 7 days in the setting of SARS-CoV-2 pneumonia treatment.

Patients who meet inclusion criteria and do not have any exclusion criteria will be randomized to receive open treatment 1:1:1

DETAILED DESCRIPTION:
Identifying treatment options is critical to the SARS-CoV-2 outbreak response. Currently there is no vaccine and treatments used are not specifically designed for this virus; They are drugs used for other pathologies. We have identified possible drugs with a known safety profile, selected the most promising ones and designed 3 combinations to select the one with the best results in clinical improvement of pneumonia due to Covid-19.

-Virus entry inhibitors: broad spectrum antivirals (antimalarials). They block viral infection by increasing endosomal pH necessary for virus / cell fusion, as well as interfering with glycosylation of cellular SARS-CoV receptors. It also has immunomodulatory activity, which can enhance antiviral effect. Latest evidence from the UK RECOVERY and WHO SOLIDARITY trials suggest that antimalarials do not provide clinical benefit in hospitalized patients with COVID-19.

Baricitinib, Janus kinase inhibitor, showing high affinity for AAK1. Disruption of AAK1 (one of the known regulators of viral endocytosis) could block passage of SARS-CoV-2 to cells and also the intracellular assembly of virus particles. Furthermore, it has the capacity to bind cyclin G-associated kinase, another regulator of endocytosis. You can limit systemic inflammatory response and cytokine production by inhibiting the JAK-STAT32 pathway.

Imatinib; Antitumor agent inhibitory activity of some tirsin kinases (TK), especially fusion oncoprotein BCR-ABL1, c-kit and native kinase ABL1. It has shown antiviral properties in early stages of infection against SARS-CoV and MERS-CoV, phylogenetically related to SARS-CoV2. In addition, it has been linked to reduced inflammation and improved endothelial barrier and pulmonary edema.

-Protease inhibitors: lopinavir / ritonavir (HIV treatment); expected interactions with SARS-CoV-2 proteases; The therapeutic effect of ritonavir and lopinavir could be mainly due to its inhibitory effect on coronavirus endopeptidase C30. The RECOVERY clinical trial investigators have also reviewed the data concluding that LPV / r does not provide clinical benefit in hospitalized patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* ≥18 years
* Confirmed diagnosis Pneumonia Covid19 + (Pneumonia confirmed radiologically and positive test for detection of SARS-CoV-2 RNA in respiratory samples)
* ECOG functional state 0 or 1
* Less than 10 days from onset of symptoms saw.
* NO contraindication for medication
* ECG QT < < 440 ms males and < 460 ms females
* Adequate liver, kidney and hematological function (or within the safety range to use these drugs):

  1. Absolute granulocyte count> 1.5 x 109 / L
  2. Absolute platelet count> 100 x 109 / L
  3. Hb> 10 g / dL
  4. Cr <1.5 mg / dL or Clearance> 50mL / min
  5. Bilirubin <3 ULN
  6. AST / ALT ≤ 2.5 times ULN

Exclusion Criteria:

* No Covid confirmation
* No pneumonia
* Previous treatment with any of the study drugs
* Concomitant serious medical condition:

  1. Congestive Heart failure
  2. Acute myocardial infarction 6 months prior
  3. Unstable Angina
  4. Cardiomyopathy
  5. Unstable Ventricular Arrhythmia
  6. Uncontrolled Hypertension
  7. Uncontrolled psychotic disorders
  8. Serious active infections
  9. HIV infections
  10. Active hepatitis
  11. Neoplasia in active cancer treatment
* Inability to take oral medication or malabsorption syndrome saw.
* Inability to comply with study and follow-up procedures
* History of only relevant thromboembolic or hemorrhagic episodes in the last 6 months
* Contraindication to any study medication
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
time to clinical improvement | baseline to day 14
  time from inclusion to improvement by 2 points on the "seven-category ordinal scale" or high, whichever comes first

SECONDARY OUTCOMES:
Safety of treatments | through study completion, an average of 1 month
  number of serious adverse effects and premature discontinuation of treatment
Tolerability of treatments | during treatment and up to 30 days after the last treatment dose
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0

OTHER OUTCOMES:
Biomarkers and genetic markers of susceptibility to SARS-CoV-2 | baseline
  Possible biomarkers and genetic markers of susceptibility to SARS-CoV-2 using high-performance techniques with serum DNA from the participants

CONTACTS AND LOCATIONS:
Overall Officials: David Bernal, Ph MD, Principal Investigator — Hospital Universitario de Fuenlabrada
Locations (1):
- Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No